CLINICAL TRIAL: NCT05715697
Title: The First Affiliated Hospital of Xinjiang Medical University
Brief Title: Renal Denervation in Patients With Chronic Heart Failure With Preserved Ejection Fraction
Acronym: RDN-HFPEF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xinjiang Medical University (Other)
Collaborators: First Affiliated Hospital of Xinjiang Medical University (Other)
Responsible Party: Principal Investigator, Xiang Xie, Head of Hypertension Department, Clinical Professor, First Affiliated Hospital of Xinjiang Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20230126-03
Record Dates: First submitted 2023-01-26; First posted 2023-02-08 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Renal Denervation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Renal denervation and maintenance of heart failure medications (Experimental): Renal denervation in patients with HFpEF and uncontrolled hypertension
  Interventions: Procedure: Renal denervation and maintenance of heart failure medications
- Sham intervention, maintenance of heart failure medications (Sham Comparator): Sham Treatment. After 1 year, cross-over is planned in all sham-treated patients and this patients will also receive a renal denervation.
  Interventions: Procedure: Sham procedure and maintenance of heart failure medications

INTERVENTIONS:
Procedure: Sham procedure and maintenance of heart failure medications — Sham intervention, maintenance of heart failure medications
  Arms: Sham intervention, maintenance of heart failure medications
Procedure: Renal denervation and maintenance of heart failure medications — Renal denervation and maintenance of heart failure medications
  Arms: Renal denervation and maintenance of heart failure medications

SUMMARY:
This study aims to explore the potential of RDN as a therapy for HFpEF in a Prospective, Multicenter, Randomized, Blinded, Sham-controlled Study.

DETAILED DESCRIPTION:
Heart failure is one of the most important diseases worldwide, with a 5-year mortality of up to 75% in symptomatic patients. While substantial progress has been made in the treatment of patients with reduced left ventricular ejection fraction (HFrEF), mortality for patients with heart failure and preserved ejection fraction (HFpEF) remains unchanged, despite a comparable prevalence and mortality of the disease as for heart failure with reduced ejection fraction. Heart failure with preserved ejection fraction has a high mortality, which is contrasted by a total absence of therapy options besides symptomatic diuretic treatment. This study aims to explore the potential of RDN as a therapy for HFpEF in a Prospective, Multicenter, Randomized, Blinded, Sham-controlled Study.

ELIGIBILITY:
Inclusion Criteria:

1. signs or symptoms of heart failure;
2. normal or mildly abnormal systolic LV function (LVEF ≥ 50%);
3. evidence of diastolic LV dysfunction.
4. Individual should fulfill the diagnostic WHO criteria for hypertension: SBP > 140 mmHg and/or DBP > 90 mmHg, and is treated with at least 2 antihypertensive drugs. This treatment is expected to be maintained for at least 6 months. Using this regimen the blood pressure should be adequately controlled (< 140/90mmHg by 24 hour ambulatory BP measurement).
5. Individual is adhering to a stable drug regimen HFNEF, with no changes for a minimum of 2 weeks prior to enrollment, and which is expected to be maintained for at least 6 months.

Exclusion Criteria:

1. Known secondary cause of hypertension
2. Anatomy not eligible for renal denervation
3. Systolic heart failure (LVEF < 50%)
4. Individual has an estimated glomerular filtration rate (eGFR) of < 30mL/min/1.73m2, using the MDRD calculation.
5. Individual has any serious medical condition, which in the opinion of the investigator, may adversely affect the safety and/or effectiveness of the participant or the study (i.e., patients with clinically significant peripheral vascular disease, abdominal aortic aneurysm, bleeding disorders such as thrombocytopenia, haemophilia, significant anaemia, or arrhythmias such as atrial fibrillation).
6. Individual is pregnant, nursing or planning to be pregnant.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline E/E' at 12 months | 12 months after treatment
  Echocardiography will be used to measure the E/E'

SECONDARY OUTCOMES:
Number of participants with adverse events | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang, China